CLINICAL TRIAL: NCT01749111
Title: Randomized Study to Compare Post Bone Marrow Transplant Cyclophosphamide With the Combination of Methotrexate Plus Calcineurin Inhibitor for Graft Versus Host Disease Prophylaxis
Brief Title: Comparison Between Cyclophosphamide and Combination of Methotrexate + Calcineurin Inhibitor for GVHD Prophylaxis
Acronym: CICLODECH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Paulo Vidal Campregher, MD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GEDECH-2012
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoid Leukemia; Myeloproliferative Disease; Myelodysplastic Syndrome; Chronic Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: bone marrow transplantation; graft versus host disease; Acute myelogenous leukemia; Acute lymphoid leukemia; Myeloproliferative disease; Myelodysplastic syndrome; Chronic myeloid leukemia; chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myeloproliferative Disorders; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Graft vs Host Disease | interventions — Cyclophosphamide; Methotrexate; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Graft versus host disease prophylaxis will be done with cyclophosphamide 50 mg/kg on day +3 and day +4
  Interventions: Drug: ARM A Cyclophosphamide
- Arm B (Active Comparator): In this arm, patients will receive a combination of methotrexate and a calcineurin inhibitor as graft versus host disease prophylaxis
  Interventions: Drug: ARM B Calcineurin inhibitor and methotrexate

INTERVENTIONS:
Drug: ARM A Cyclophosphamide — Cyclophosphamide 50 mg/kg on day+3 and day+4 after bone marrow transplantation
  Other Names: Cyclophosphamide
  Arms: Arm A
Drug: ARM B Calcineurin inhibitor and methotrexate — Graft versus host disease prophylaxis will be done with the combination of a calcineurin inhibitor (either tacrolimus or cyclosporine) and methotrexate
  Other Names: Calcineurin inhibitor and methotrexate
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine whether cyclophosphamide post bone marrow transplant increases the rate of patients alive, in remission and without immunosuppression, one year after transplant, when compared with the combination of methotrexate and calcineurin inhibitor

DETAILED DESCRIPTION:
We propose a study in which 150 patients will receive graft versus host disease prophylaxis with cyclophosphamide 50 mg/kg on day +3 and day +4 after bone marrow transplantation, and 150 patients will receive the usual combination of methotrexate and calcineurin inhibitor. The study was designed to last for 4 years. The primary endpoint is the rate of patients alive, in remission and without immunosuppression, one year after transplant. The assignment for each arm of the study will be done through simple randomization.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 to 60 years of age.
* The patient should have a HLA matched donor
* The patient must need a bone marrow transplant for a malignant disease (Acute leukemia, myelodysplastic syndrome, myeloproliferative disease or myelodysplastic/myeloproliferative disease)
* Patients want to participate in the study, and able to give informed consent.

Exclusion Criteria:

* Previous auto o allogeneic hematopoietic stem cell transplant
* Performance Status >2 (ECOG).
* Pregnancy
* HIV positive
* Active Infection
* Cardiac disease with ejection fraction < 45%
* Lung disease with FEV1, FVC ou DLCO <50% of predicted values.
* Renal Insufficiency with creatinine clearance < 60 ml/minute.
* Liver disease with bilirubin levels > twice the reference value or ALT or AST > three times the normal reference.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The rate of patients alive, in remission and without immunosuppression, one year after bone marrow transplantation. | one year
  The rate of patients alive, in remission and without immunosuppression, one year after bone marrow transplantation.

SECONDARY OUTCOMES:
Cumulative incidence of chronic graft versus host disease, one year after bone marrow transplantation | one year
  Cumulative incidence of chronic graft versus host disease, one year after bone marrow transplantation

OTHER OUTCOMES:
Cumulative incidence of disease relapse, one year after bone marrow transplantation | one year
  Cumulative incidence of disease relapse, one year after bone marrow transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Paulo V Campregher, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein 's (IIEP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Luznik L, Bolanos-Meade J, Zahurak M, Chen AR, Smith BD, Brodsky R, Huff CA, Borrello I, Matsui W, Powell JD, Kasamon Y, Goodman SN, Hess A, Levitsky HI, Ambinder RF, Jones RJ, Fuchs EJ. High-dose cyclophosphamide as single-agent, short-course prophylaxis of graft-versus-host disease. Blood. 2010 Apr 22;115(16):3224-30. doi: 10.1182/blood-2009-11-251595. Epub 2010 Feb 2. PMID 20124511